CLINICAL TRIAL: NCT02002949
Title: Cost-Utility of Conventional Hemodialysis (CHD) Vs Short Daily Hemodialysis (SDHD) for Patients Coming From Peritoneal Dialysis (HAPD/CAPD): A Randomized Controlled Trial
Brief Title: Conventional Hemodialysis Vs Short Daily Hemodialysis for Patients Coming From Peritoneal Dialysis (HAPD/CAPD)
Acronym: CHDvsSDHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Responsible Party: Principal Investigator, Loreto GESUALDO, FULL PROFESSOR, Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: RF-2010-2314193
Record Dates: First submitted 2013-11-20; First posted 2013-12-06 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: End Stage Renal Disease
Keywords: Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Short daily hemodialsysis (Experimental): Short Daily Hemodialysis (SDHD) - 5 or 6 treatments per week for approximately 3 hours (range 2 to 4 hours) per treatment, to be performed at the patient's home, using any hemodialysis machine as chosen by the responsible clinician in each participating center
  Interventions: Procedure: Short daily hemodialysis
- Conventional hemodialysis (Active Comparator): Conventional Hemodialysis (CHD) - 3 treatments per week for approximately 4 hours (range 3 hours and 30 minutes to 4 hours) per treatment, to be performed in a dialysis clinic using any hemodialysis machine as chosen by the responsible clinicians in each participating center
  Interventions: Procedure: Conventional hemodialysis

INTERVENTIONS:
Procedure: Short daily hemodialysis — 5 or 6 treatments per week for approximately 3 hours (range 2 to 4 hours) per treatment, to be performed at the patient's home, using any hemodialysis machine as chosen by the responsible clinician in each participating center
  Arms: Short daily hemodialsysis
Procedure: Conventional hemodialysis — 3 treatments per week for approximately 4 hours (range 3 hours and 30 minutes to 4 hours) per treatment, to be performed in a dialysis clinic using any hemodialysis machine as chosen by the responsible clinicians in each participating center
  Arms: Conventional hemodialysis

SUMMARY:
The purpose of this randomized study is to determine if the home SDHD is a suitable alternative to conventional dialysis performed in a dialysis center for patients suffering from chronic kidney disease from Peritoneal Dialysis (HAPD/CAPD).

The adequacy of this alternative dialysis technique confirms that the SDHD at home is a viable option for patients coming from HAPD/CAPD and indeed support the clinical benefits of home SDHD compared with those of conventional dialysis: lowering blood pressure and lower use of antihypertensive drugs , improving the quality of life, maintenance of residual renal function related to a reduced risk of death and reduction in operating costs of dialysis and patient transport.

DETAILED DESCRIPTION:
Conventional Hemodialysis - 3 treatments per week for approximately 4 hours- will be performed in a dialysis clinic using any hemodialysis machine. Short Daily Hemodialysis - 5 or 6 treatments per week for approximately 2-4 hours per treatment- will be performed in the patient's home, using any hemodialysis machine. Partecipants randomized to SDHD will undergo an intensive home hemodialysis training program expected to take 2-6 weeks to complete. Qualified healthcare professionals will train each SDHD subject's partner to perform dialysis using any hemodialysis machine as chosen by clinicians. At baseline visit, before the first study treatment in either the SDHD or CHD arm, the following data will be collected: demographic information, ESRD history, EuroQol EQ-5D-5L questionnaire, vital sign, blood laboratory test results, KT/V parameters, 24 hour timed urine collection test results, comorbid conditions, vascular access type, current medications. After hemodialysis start, patients will be followed up to 12 months with data collection at 1,3,6 and 12 months. At each visit, the following data will be collected: EuroQol EQ-5D-5L questionnaire, vital sign, blood laboratory test results, KT/V parameters, 24 hour timed urine collection test results, adverse events, vascular access type, current medications. During this study, the following parameters will be strictly monitored: treatment costs, medications, number of hospitalization admissions, number of days in hospital and reasons for hospitalizations, additional costs informations.

Home hemodialysis could be an integrated therapeutic option favoring the de-hospitalization of patients requiring hemodialysis. Aim of this study is to offer the patient a better quality of life, to create the conditions for an improvement in blood pressure, phosphate control, of cardiovascular morbidity and mortality, and to reduce costs for the National Health Service.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of end-stage renal disease
2. Currently performing Peritoneal Dialysis (HAPD and CAPD) for a minimum of 3 months.
3. Age 18 years or older.
4. Suitability for SDHD, determined on the basis of the following conditions:

   * willingness to be trained and perform frequent hemodialysis at home;
   * physically and mentally capable of performing frequent hemodialysis at home;
   * evaluation of the subject's home environment by a physician, training nurse and /or social worker;
   * a home dialysis partner willing to assist the participant in performing treatments at home;
   * agreement by a multidisciplinary (physician, nurse and any other professionals) team that the subject is suitable for SDHD.
5. Expected survival of at least one year.
6. Ability to understand and willingness to sign an informed consent statement.

Exclusion Criteria:

1. Current enrollment in another investigational drug or device trial which might impact the outcomes measures planned in this study.
2. Being scheduled for change of modality or plans to relocate to an area outside of the clinical center.
3. Cancer
4. Pregnancy-lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
mean quality-adjusted life year (QALY) score in the first year after the start of dialysis | one year

SECONDARY OUTCOMES:
dialysis related cost of care | one year
transportation costs per patient per year for the journeys "home-hospital-home" | one year
ratio nurse/patients | one year
hospitalization rate (admissions and days | one year
weekly standardized Kt/V delivered | one year
systolic blood pressure and use of antihypertensive medications | one year
  blood pressure will be assessed for a year and measured in mmHg. It will be evaluated if the patient will need to increase the antihypertensive therapy or to reduce it
mineral metabolism, anemia parameters and nutritional parameters | one year
  As of mineral metabolism, it will be assessed serum calcium levels (expressed in mg per deciliter), serum phosphorus levels (expressed in mg per deciliter), parathormone levels (expressed in pg/ml). As of anemia, it will evaluated hemoglobin levels (expressed in g per deciliter), hematocrit (expressed in %), serum ferritin (μg/l) , transferrin saturation (expressed in %). Albumin (g/dl) will be a nutritional parameter
maintenance of residual renal function | one year
  it will be assessed residual diuresis per day expressed in ml and residual creatinine clearance expressed in ml/min

CONTACTS AND LOCATIONS:
Overall Officials: Loreto LG GESUALDO, MD, Principal Investigator — AOUConsorziale, Bari, Italy
Locations (31):
- Italy (31):
  - AUO Policlinico Consorziale, Bari, BA
  - Ospedale Santa Marta e Santa Venera di Acireale, Acireale
  - A.O.U. Ospedali Riuniti di Ancona, Ancona
  - Presidio Ospedaliero 1 - Arezzo, "San Donato", Arezzo
  - Policlinico Universitario S. Orsola-Malpighi, Bologna
  - Azienda Ospedaliera G. Brotzu, Cagliari
  - Ospedale S. Giacomo Apostolo, Castelfranco Veneto
  - Ospedale per l'emergenza Cannizzaro Catania, Catania
  - Ospedale SS.Annunziata, Chieti
  - Ospedale Civile di Cremona, Cremona
  - Azienda Ospedaliero Universitaria "OO.RR." di Foggia, Foggia
  - ASL 12 Di Viareggio - Ospedale Versilia, Lido di Camaiore
  - Seconda Università degli Studi di Napoli, Napoli
  - Secondo Policlinico-Azienda Ospedaliera Universitaria "Federico II", Napoli
  - Secondo Ospedale S. Francesco, ASL 3 S, Nuoro
  - Ospedale Civile Spirito Santo, Pescara
  - Ospedale Civile di Piacenza, Piacenza
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Ospedale G. B. Grassi, Roma
  - Università Cattolica Del Sacro Cuore, Roma
  - Ospedale Santa Maria della Misericordia, Rovigo
  - Ospedale D. Anna, San Fermo della Battaglia
  - Ospedale Civile San Giovanni Di Dio, San Michele
  - Ospedale Principe di Piemonte, Senigallia
  - Ospedale Umberto I di Siracusa, Syracuse
  - Ospedale Mazzini, Teramo
  - Ospedale San giovanni Battista Molinette, Torino
  - Ospedale San giovanni Bosco, Torino
  - Ospedale Santa Chiara, Trento
  - Ospedale Treviglio - Caravaggio, Treviglio
  - Ospedale Civile di Voghera, Voghera